CLINICAL TRIAL: NCT07075679
Title: Use of Artificial Intelligence in Breast Cancer Screening: Impact of AI-Assisted Single Reading by One Radiologist on Screening Quality Indicators Compared to Standard Double Reading by Two Radiologists Without AI
Brief Title: Screening Mammography: Single Reading by One Radiologist With AI vs. Double Reading by Two Radiologists (AI-BCSQ)
Acronym: AI-BCSQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 03062025; IGA_LF_2024_022 (Other Grant/Funding Number: Internal Grant of the Palacky University)
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Screening; Artificial Intelligence (AI); Breast Cancer Screening and Diagnosis
Keywords: breast cancer; screening; artificial intelligence
MeSH Terms: conditions — Disease; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with AI (Experimental): Asymptomatic women aged 45-69 participating in breast cancer screening programme, reading of mammograms by one radiologist with AI support.
  Interventions: Diagnostic Test: Group with AI iCAD version 3
- Group without AI (Other): Asymptomatic women aged 45-69 participating in breast cancer screening programme, reading of mammograms by two radiologists without AI (current practice).
  Interventions: Diagnostic Test: Group without AI

INTERVENTIONS:
Diagnostic Test: Group with AI iCAD version 3 — Reading mammograms by one radiologist with AI support
  Arms: Group with AI
Diagnostic Test: Group without AI — Standard double reading by two radiologists without AI.
  Arms: Group without AI

SUMMARY:
A randomized prospective study comparing the evaluation of mammography images in a breast cancer screening programme by a single radiologist with AI support versus standard double reading by two radiologists without AI support.

DETAILED DESCRIPTION:
In the intervention group, the first reading of the screening mammogram will be performed by one radiologist with AI support. After this AI-assisted first reading is completed and recorded for the study, a standard second reading will be carried out by another radiologist. This ensures that the legal requirement for double reading in the breast cancer screening program is maintained.

In the control group, mammograms will be evaluated according to the current standard practice - that is, independently by two radiologists without AI support.

Participants will be divided to the two groups based on a randomization scheme that determines specific days for evaluation with AI (Group 1) and without AI (Group 2). The randomization ensures equal distribution of weekdays between the two groups to minimize bias due to variability in daily workflow, diagnostic/screening ratios, or other operational factors.

ELIGIBILITY:
Inclusion Criteria:

* age 45-69, asymptomatic woman participating in breast cancer screening programme

Exclusion Criteria:

* clinical signs of breast disease - indication for diagnostic mammography

Ages: 45 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2028-08-03 (Estimated); Study Completion 2028-08-03 (Estimated)

PRIMARY OUTCOMES:
Further assessment rate | up to 190 days after screening mammmography
  The proportion of women udergoing follow-up examinations within 0-190 days after screening mammography.

SECONDARY OUTCOMES:
Cancer Detection Rate | up to 1 year after screening mammography
  The number of cancers detected per 1,000 women screened.
Recall Rate | up to 190 days after screening mammography
  The proportion of women recalled for follow-up examinations withing 1-190 days after screening mammography.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsen M, Olstad CF, Lee CI, Hovda T, Hoff SR, Martiniussen MA, Mikalsen KO, Lund-Hanssen H, Solli HS, Silberhorn M, Sulheim AO, Auensen S, Nygard JF, Hofvind S. Performance of an Artificial Intelligence System for Breast Cancer Detection on Screening Mammograms from BreastScreen Norway. Radiol Artif Intell. 2024 May;6(3):e230375. doi: 10.1148/ryai.230375. PMID 38597784
- [Result] Lambin P, Leijenaar RTH, Deist TM, Peerlings J, de Jong EEC, van Timmeren J, Sanduleanu S, Larue RTHM, Even AJG, Jochems A, van Wijk Y, Woodruff H, van Soest J, Lustberg T, Roelofs E, van Elmpt W, Dekker A, Mottaghy FM, Wildberger JE, Walsh S. Radiomics: the bridge between medical imaging and personalized medicine. Nat Rev Clin Oncol. 2017 Dec;14(12):749-762. doi: 10.1038/nrclinonc.2017.141. Epub 2017 Oct 4. PMID 28975929
- [Result] Tudos Z, Veverkova L, Baxa J, Hartmann I, Ctvrtlik F. The current and upcoming era of radiomics in phaeochromocytoma and paraganglioma. Best Pract Res Clin Endocrinol Metab. 2025 Jan;39(1):101923. doi: 10.1016/j.beem.2024.101923. Epub 2024 Aug 23. PMID 39227277
- [Result] McDonald ES, Conant EF. Can AI Reduce the Harms of Screening Mammography? Radiol Artif Intell. 2023 Oct 25;5(6):e230304. doi: 10.1148/ryai.230304. eCollection 2023 Nov. No abstract available. PMID 38074781
- [Result] Letter H, Peratikos M, Toledano A, Hoffmeister J, Nishikawa R, Conant E, Shisler J, Maimone S, Diaz de Villegas H. Use of Artificial Intelligence for Digital Breast Tomosynthesis Screening: A Preliminary Real-world Experience. J Breast Imaging. 2023 May 22;5(3):258-266. doi: 10.1093/jbi/wbad015. PMID 38416890
- [Result] Dahlblom V, Dustler M, Tingberg A, Zackrisson S. Breast cancer screening with digital breast tomosynthesis: comparison of different reading strategies implementing artificial intelligence. Eur Radiol. 2023 May;33(5):3754-3765. doi: 10.1007/s00330-022-09316-y. Epub 2022 Dec 11. PMID 36502459
- [Result] Eisemann N, Bunk S, Mukama T, Baltus H, Elsner SA, Gomille T, Hecht G, Heywang-Kobrunner S, Rathmann R, Siegmann-Luz K, Tollner T, Vomweg TW, Leibig C, Katalinic A. Nationwide real-world implementation of AI for cancer detection in population-based mammography screening. Nat Med. 2025 Mar;31(3):917-924. doi: 10.1038/s41591-024-03408-6. Epub 2025 Jan 7. PMID 39775040
- [Result] Diaz O, Rodriguez-Ruiz A, Sechopoulos I. Artificial Intelligence for breast cancer detection: Technology, challenges, and prospects. Eur J Radiol. 2024 Jun;175:111457. doi: 10.1016/j.ejrad.2024.111457. Epub 2024 Apr 16. PMID 38640824
- [Result] Lang K, Dustler M, Dahlblom V, Akesson A, Andersson I, Zackrisson S. Identifying normal mammograms in a large screening population using artificial intelligence. Eur Radiol. 2021 Mar;31(3):1687-1692. doi: 10.1007/s00330-020-07165-1. Epub 2020 Sep 2. PMID 32876835
- [Result] Lang K, Josefsson V, Larsson AM, Larsson S, Hogberg C, Sartor H, Hofvind S, Andersson I, Rosso A. Artificial intelligence-supported screen reading versus standard double reading in the Mammography Screening with Artificial Intelligence trial (MASAI): a clinical safety analysis of a randomised, controlled, non-inferiority, single-blinded, screening accuracy study. Lancet Oncol. 2023 Aug;24(8):936-944. doi: 10.1016/S1470-2045(23)00298-X. PMID 37541274
- [Result] Dembrower K, Crippa A, Colon E, Eklund M, Strand F; ScreenTrustCAD Trial Consortium. Artificial intelligence for breast cancer detection in screening mammography in Sweden: a prospective, population-based, paired-reader, non-inferiority study. Lancet Digit Health. 2023 Oct;5(10):e703-e711. doi: 10.1016/S2589-7500(23)00153-X. Epub 2023 Sep 8. PMID 37690911
- [Result] Chang YW, Ryu JK, An JK, Choi N, Park YM, Ko KH, Han K. Artificial intelligence for breast cancer screening in mammography (AI-STREAM): preliminary analysis of a prospective multicenter cohort study. Nat Commun. 2025 Mar 6;16(1):2248. doi: 10.1038/s41467-025-57469-3. PMID 40050619
- See also: 1. European Commission: Joint Research Centre, ECIBC at a Glance - European Commission Initiative on Breast Cancer, Publications Office of the European Union, 2023 — https://data.europa.eu/doi/10.2760/908946